CLINICAL TRIAL: NCT06944288
Title: Microbiota as Early Diagnostic and predictivE Factor for Osteoarthritic Degeneration and Microbial Contamination (MILESTONE)
Brief Title: Microbiota as Early Diagnostic and predictivE Factor for Osteoarthritic Degeneration and Microbial Contamination
Acronym: MILESTONE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Azienda Ospedaliera di Rilievo Nazionale A.Cardarelli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12377976
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Knee Prosthesis; Knee Prosthesis Infection; Disbiosis
MeSH Terms: conditions — Dysbiosis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Prosthesis surgery Revision of infected prosthesis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SURGERY (Other): TOTAL KNEE REPLACEMENT SURGERY AND REVISION SURGERY OF INFECTED KNEE PROSTHESIS
  Interventions: Procedure: total knee replacement

INTERVENTIONS:
Procedure: total knee replacement — The Orthopedic Surgeon will remove the damaged cartilage and bone then implant the new metal and plastic knee to restore the alignment and function of your knee. The surgical procedure takes about 1-2 hours on average. While in case of infection, an antibiotic cement is inserted, which will be removed with the subsequent prosthetic implant surgery. Finally, prosthetic components can be more filling, depending on the amount of bone that is previously removed.

SUMMARY:
The patient(s) will participate in a clinical study that aims to investigate how the gut microbiota may influence the proper functioning of joints in the body and how it may affect the development of early osteoarthritis (OA), periprosthetic joint infection (PJI), and recovery after total joint replacement.

In particular, the prevalence of early OA among patients with gut dysbiosis will be studied (Objective 1). The aim is to identify gut dysbiosis as a potential diagnostic factor for early OA. The study will analyze knee MRI scans and shoulder ultrasound images of 40 patients without musculoskeletal symptoms but with confirmed gut dysbiosis.In addition, the intra-articular microbiota in 50 patients undergoing total knee replacement will be investigated. Serum LPS levels during surgery and fecal microbiota before surgery and during postoperative recovery will be assessed (Objective 2). Postoperative recovery will be assessed based on criteria such as time off crutches and subjective scores.

Finally, this will explore the correlation between gut microbiota and contaminating germs in periprosthetic infections. (Objective 3). 40 patients undergoing joint revision surgery for septic failure of a knee or hip replacement and 40 patients undergoing revision surgery for aseptic loosening for PJI will undergo gut microbiota analysis. Comparison between the two groups will allow evaluation of whether PJI causes changes in the gut microbiota.

The patients will be included in the study under

* objective 1
* objective 2
* objective 3

DETAILED DESCRIPTION:
The study is a multicentre observational study divided into 3 objectives:

Objective #1 is to enrol 40 patients with established intestinal dysbiosis and no musculoskeletal symptoms. Patients with potential dysbiosis will undergo an initial (V1) gastroenterological examination at the Operative Unit of Gastroenterology and Digestive Endoscopy in Humanitas, where they will be asked to join the clinical study. Each patient will be explained the study through the means of the informed consent process, and those who wish to join the study will sign the informed consent form. For each patient, the Bristol scale will be used as a tool to categorize the patients' stool as reported by the patient; a stool sample collection kit will be provided to the patient together with its instructions for use. Patients will be instructed to provide a stool sample (V2) at the immunology and microbiota unit laboratory. On the same occasion, the clinician will perform a buccal swab to collect a saliva sample from the patient (see section 8 for specifics). Both samples will initially be stored at the Biobank - Cancer Center (Istituto Clinico Humanitas - Via Manzoni 56, 20089 Rozzano (MI)) under the responsibility of Dr. Daniela Pistillo and will then be processed at the laboratory of the immunology and microbiota unit and will be used for confirming the dysbiosis diagnosis. If the patient is not positive for dysbiosis markers, he/she will be classified as SCREENING FAILURE; if the dysbiosis is confirmed, the patient will be asked to come to another visit (V3) where he/she will undergo a MRI of the knee and a shoulder ultrasound scan in order to check for early osteoarthritis signs. Optional orthopaedic examination may be performed. Blood test will also be performed part of the samples of which will be used to evaluate biomarkers and will initially be stored at the Biobank - Cancer Center (Istituto Clinico Humanitas - Via Manzoni 56, 20089 Rozzano (MI)) with Dr. Daniela Pistillo in charge and will subsequently be processed. The other part of the blood samples on which insulin, glycated haemoglobin and glucose will be analysed will be sent to the Central Analysis Laboratory within ICH (see section 8 for details).

Objective #2 is to enrol 50 patients undergoing total knee arthroplasty (TKA). Patients scheduled to undergo TKA will undergo a pre-hospitalization orthopaedic examination (V1) where he/she will be informed about the clinical study. If he/she agrees to join the study, he/she will sign the informed consent form and will follow study procedures: questionnaires will be administered and the patient will receive a stool sample collection kit together with its instructions for use. The stool sample will be used for DNA extraction at the immunology and microbiota unit laboratory and subsequent metagenomic analysis. Patient will be instructed to hand over the stool sample during hospital visit for TKA (V2), during which intra-articular tissue samples will be collected for metagenomics. In addition, buccal swab and blood samples of the patient undergoing the surgery will be collected before surgery. Saliva, stool and blood samples for biomarkers will initially be stored at the Biobank - Cancer Center (Istituto Clinico Humanitas - Via Manzoni 56, 20089 Rozzano (MI)) under the responsibility of Dr. Daniela Pistillo and will subsequently be processed at the laboratory of the immunology and microbiota unit. The other part of the blood samples on which insulin, glycated haemoglobin and glucose will be analysed will be sent to the ICH's in-house Central Analysis Laboratory. On discharge, patient will be provided another stool collection kit. One month after surgery (V3), a follow-up examination will be performed, where patient will bring the second stool sample and will undergo another buccal swab which will also be analysed by the same laboratory (see section 8). For stool and saliva samples of V3, the storage and analysis procedure is the same as for V2. In addition, the patient will fill in the KSS questionnaires.

Objective #3 involves the enrolment of 80 patients undergoing joint revision surgery who are further divided into:

Group 1: 40 patients for septic failure of a knee or hip replacement. Group 2: 40 patients for aseptic loosening for PJI Patients will undergo a pre-hospitalization visit (V1) with orthopaedic check-up, where they will be asked to join the clinical study. Each patient will be explained the study through the means of the informed consent process, and those who wish to join the study will sign the informed consent form. Patient will be provided a stool sample collection kit for DNA extraction at the immunology and microbiota unit laboratory and subsequent metagenomic analysis. The patient will be instructed to hand over the stool sample during hospital visit for revision surgery (V2) (see section 8).

ELIGIBILITY:
Inclusion Criteria:

* proven gut dysbiosis (increased Firmicutes/Bacteroidetes (F/B) phyla ratio and increased permeability); age range 18-50 years old.
* patients undergoing total knee replacement surgery
* patients undergoing joint revision surgery for septic failure of a knee or hip prostheses; patients undergoing revision surgery for aseptic mobilization for PJI

Exclusion Criteria:

* musculoskeletal symptoms; previous shoulder or knee surgery; previous shoulder or knee known pathological conditions; rheumatological diseases
* any concurrent or previous diseases or conditions which might negatively affect the surgery
* major predisposing factor for gut dysbiosis (antibiotic therapy in the last 6 months, BMI > 40 and inflammatory bowel disease); chronic inflammatory joint diseases (e.g., rheumatoid arthritis, psoriatic arthritis); acute (< 90 days after the index procedure) and late hematogenous (symptoms of less than three weeks duration) infections; an inadequate amount of synovial fluid (< 10 mL) for culture, WBC, and PMN (neutrophil) percentage determinations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 : to identify gut dysbiosis as a potential diagnostic tool for early OA. | 1 year
  The study aims to establish gut dysbiosis as a potential diagnostic tool for early OA. If a strong association between gut dysbiosis and early OA is found, it could contribute to the development of a diagnostic protocol for early OA. The identification of gut dysbiosis as an early marker of OA could represent an additional diagnostic tool, allowing for early intervention and prevention of further progression of the disease. Early recognition of OA would allow a precocious and timely intervention which could positibely alter the natural history of this condition.
Outcome 2: to investigate the intraarticular microbiota, serum LPS levels during surgery, and fecal microbiota before surgery and during recovery. | 1 year
  The analysis may reveal specific microbial imbalances or dysregulated pathways in the gut microbiota and serum LPS levels that are correlated with post-operative recovery outcomes. The study seeks to determine whether there is a correlation between the gut microbiota composition and post-operative recovery after total kneereplacement (TKA). It is expected that certain microbial taxa or functional pathways i n the gut microbiota will be associated with faster recovery, as indicated by shorter time taken to abandon crutches and higher subjective scores (e.g., KneeSociety Score, KSS score). The study aims to investigate the role of the gut microbiota as a predicting factor for joint arthroplasty recovery. If a significant correlation is found between specific microbial imbalances or dysregulated pathways and post-operative recovery outcomes, it could indicate that the gut microbiota can serve as a predictive factor for recoveryafter TKA.
Outcome 3: to investigate if periprosthetic joint infections (PJI) influences gut microbiota environment predisposing to gut dysbiosis, which negatively affects life expectancy in these patients. | 1 year
  The analysis may reveal specific microbial imbalances or dysregulated pathways in the gut microbiota that are correlated with the presence of PJI. It is expected that patients with PJI will exhibit distinct alterations in the gut microbiota compared to patients undergoing revision surgery for aseptic mobilization. The analysis may establish a correlation between specific microbial taxa or functional pathways in the gut microbiota and the occurrence of PJI.

CONTACTS AND LOCATIONS:
Overall Officials: TOMMASO BONANZINGA, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT06944288/Prot_SAP_000.pdf